CLINICAL TRIAL: NCT00574054
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation Treatment for Dementia and Other Related Mental Illness.
Brief Title: Far Infrared Radiation Treatment of Dementia and Other Mental Illness
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder & President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-DEM-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Dementia
Keywords: Familial Dementia; Semantic Dementia; Senile Paranoid Dementia
MeSH Terms: conditions — Dementia; Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Radiation: Far Infrared

INTERVENTIONS:
Radiation: Far Infrared — Far infrared radiation (5 μm to 20 μm wavelength) for 30 to 40 minutes per treatment session.

SUMMARY:
This trial is a preliminary study to determine the use of far infrared radiation for the treatment of dementia and other mental sickness.

DETAILED DESCRIPTION:
Dementia is the progressive decline in cognitive function due to damage or disease in the brain beyond what might be expected from normal aging. Particularly affected areas include memory, attention, language, and problem solving. Especially in the later stages of the condition, affected persons may be disoriented in place and in person (not knowing who they are).

The prevalence of dementia is rising as the global life expectancy is rising. Particularly in Western countries, there is increasing concern about the economic impact that dementia will have in future, older populaces.

It is a disease that is strongly associated with age; 1% of those aged 60-65, 6% of those aged 75-79, and 45% of those aged 95 or older suffer from the disease.

We are postulating that the use of far infrared radiation on the central nervous system, the endocrine system and the viscera will have a positive effect on treating dementia and other neurological illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Persons age 2 or older, with dementia, Alzheimer's, Huntington's disease, Parkinson's disease, Down's syndrome, multiple sclerosis or stroke

Exclusion Criteria:

* Persons with severe mental illness that are confined to mental hospitals etc., as defined by the USA Diagnostic and Statistical Manual of Mental Disorders (DSM)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation on dementia. | 1 year

SECONDARY OUTCOMES:
The secondary end point of the study is to evaluate the therapeutic effects of far infrared radiation on other related mental illness including Alzheimer's, multiple sclerosis and stroke rehabilitation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kwasi Donyina, Ph.D., Principal Investigator — GAAD Medical Research Institute Inc.; Ken Nedd, M.D., Study Director — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada